CLINICAL TRIAL: NCT00613899
Title: Feasibility of Telesurveillance and Home Cough Assistance for Amyotrophic Lateral Patients (ALS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Michele Vitacca, Principal Investigator, Fondazione Salvatore Maugeri
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N°83_researchbookFSM2006
Record Dates: First submitted 2008-01-17; First posted 2008-02-13 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2011-07

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: home care; home rehabilitation; telemedicine; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Telesurveillance (Other): At time of discharge from hospital, 40 ALS patients willbe enrolled in a telesurveillance program (TP) for the management of cought at home.
  Two hours of an in-hospital educational training will be provided to patients and caregivers on the use of:
  1. air stacking with Ambu balloon
  2. manual manoeuvres and
  3. in-Exoflator device indications and use
  Interventions: Other: telesurveillance

INTERVENTIONS:
Other: telesurveillance — A telesurveillance program for cough assistance will be approched by the use of an in-exoflator device. Measurement of oxygen saturation (SpO2) will be performed by a Nonin 9500 oxymeter (Minneapolis Plymouth USA).
  Other Names: telemedicine

SUMMARY:
The investigators want to test feasibility of a structured program of telesurveillance and home cough assistance for ALS patients.

DETAILED DESCRIPTION:
Background: Amyotrophic Lateral Sclerosis (ALS) patients present reduction in the inspiratory and expiratory muscle strength, frequent secretions increase, insufficient expectoration ability with inevitable risk of acute respiratory failure (ARF) and necessity of hospitalizations. Recently, new mechanical tools (In-Exoflator EmersonR) are available in our hospital to help patients to expectorate during ARF. It is well noted these patients are particularly reluctant to be hospitalized to avoid further worsening in their quality of life.

Aim: the investigators want to test feasibility of a structured program of telesurveillance and home cough assistance for ALS patients.

Methods: A telesurveillance program (TP), a pulsed saturimetric device, 2 hours educational hospital sections (air stacking with Ambu balloon, manual manoeuvres and In-Exoflator indications and use) will be offered to all ALS consecutive patients.

In details the TP is structured as follows: 1) Domiciliary Telesurveillance by only one 24-h Service Centre (SC) for enrolled pts with ALS in hospital discharge phase, 2) Patients - taken care of five days/week by a nurse-tutor (NT) and respiratory therapist (RT) according to a predefined appointments, 3) for 24-hr. duration (in case of symptoms) patients can call SC and talk to pneumologists that can intervene whenever needed for diagnostic-therapeutic adjustments. 4) In case of need the patient can contact the neurologist or psychologist; 5) The RT in accordance with pneumologist can decide for a domiciliary visit to patient.

Home RT accesses and In-Exoflator activation will be prescribed when patients will present worsening of three points in pSaTO2, 30% in peak cough expiratory flow (PCEF), lack of cough ability with increase in secretions and or suctions necessity (in tracheotomy patients) and clinical symptoms (dyspnoea, fever, headache, somnolence).

Number of In-Ex and air stacking activations, ARF episodes, hospital accesses, antibiotic therapy, customer satisfaction, PCF/PEF, MIC-VC, respiratory function (MIP, MEP, FEV1, FVC, FEV1/FVC, ABG), dyspnoea (Borg scale), general disability (Hoevelaken scale and ALS Functional Rating Scale) and survival will be collected.

Expected results: 30 ALS patients (VC < 80% and 40% with tracheotomy) will be enrolled after discharge from Respiratory or Neurological units of S. Maugeri Foundation. This study will allow:

1. To test a possible alternative of care for ALS patients
2. To check patients and caregivers' acceptance
3. To measure time consuming for care team
4. To quantify patient's comfort
5. To test costs/effectiveness ratio.

ELIGIBILITY:
Inclusion criteria:

* 40 ALS patients (VC < 80% with or without tracheostomy)will be enrolled after discharge from Respiratory or Neurological units of S. Maugeri Foundation.

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2008-03 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To test a possible alternative of care for ALS patients (home vs hospital) | 6-12 months

SECONDARY OUTCOMES:
To check patients and caregivers' acceptance | 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: michele vitacca, MD, Study Chair — FSM IRCCS Lumezzane; michele vitacca, MD, Principal Investigator — FSM IRCCS LUmezzane (BS) ITALY
Locations (1):
- Michele Vitacca, Lumezzane, BS, Italy

REFERENCES:
- [Background] Sancho J, Servera E, Diaz J, Marin J. Efficacy of mechanical insufflation-exsufflation in medically stable patients with amyotrophic lateral sclerosis. Chest. 2004 Apr;125(4):1400-5. doi: 10.1378/chest.125.4.1400. PMID 15078752
- [Result] Vitacca M, Paneroni M, Trainini D, Bianchi L, Assoni G, Saleri M, Gile S, Winck JC, Goncalves MR. At home and on demand mechanical cough assistance program for patients with amyotrophic lateral sclerosis. Am J Phys Med Rehabil. 2010 May;89(5):401-6. doi: 10.1097/PHM.0b013e3181d89760. PMID 20407305
- [Derived] Paneroni M, Trainini D, Winck JC, Vitacca M. Pilot study for home monitoring of cough capacity in amyotrophic lateral sclerosis: A case series. Rev Port Pneumol. 2014 Jul-Aug;20(4):181-7. doi: 10.1016/j.rppneu.2013.11.003. Epub 2014 Feb 1. PMID 24491372
- See also: association of amyotrophic lateral sclerosis patients — http://www.aisla.it